CLINICAL TRIAL: NCT07095855
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled and Open-Label Extension Phase III Study to Evaluate the Efficacy and Safety of ZM-H1505R (Canocapavir) in Combination With Nucleos(t)Ide Analog(NAs) Compared With NAs Monotherapy in Patients With Chronic Hepatitis B Who Have Received NAs Monotherapy for at Least 12 Months
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of ZM-H1505R in Patients With CHB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZM-H1505R-301
Record Dates: First submitted 2025-07-14; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B
Keywords: ZM-H1505R; Hepatitis B; CHB
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A:ZM-H1505R + NAs (Experimental): ZM-H1505R 100mg,QD + NAs(ETV or TDF or TAF or TMF)
  Interventions: Drug: ZM-H1505R 100mg; Combination Product: NAs （"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"or"TMF"） treatments
- Group B: ZM-H1505R Placebo + NAs (Placebo Comparator): ZM-H1505R Placebo 100mg,QD + NAs(ETV or TDF or TAF or TMF)
  Interventions: Other: ZM-H1505R Placebo; Combination Product: NAs （"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"or"TMF"） treatments

INTERVENTIONS:
Drug: ZM-H1505R 100mg — ZM-H1505R(100mg,QD) will be used in Part A double-blind treatment period for 48 weeks and Part B open-label extension period 144 weeks.
  Arms: Group A:ZM-H1505R + NAs
Other: ZM-H1505R Placebo — ZM-H1505R Placebo(100mg,QD) will be used in Part A double-blind treatment period for 48 weeks.
  Arms: Group B: ZM-H1505R Placebo + NAs
Combination Product: NAs （"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"or"TMF"） treatments — All eligible subjects will be use NAs （"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"or"TMF"） treatments during the study for 148 weeks, including Part A and Part B.
  Subjects will continue to use the NAs as combination therapy before enrollment, the dosage will not be adjusted during the study. Subjects use in accordance with medical advice andinstructions.

SUMMARY:
This study is divided into two parts. Part A is a multicenter, randomized, double-blind, placebo controlled phase Ill clinical trial, designed to evaluate the efficacy and safety of ZM-H1505R in combination with NAs versus NAs monotherapy with HBV DNA ≥ 50 IU/mL and are HBeAg positive who have received NAs monotherapy for at least 12months.Part B is an open-label extension and follow-up period designed to evaluate the long-term safety and efficacy of ZM-H1505R in combination with NAs.

DETAILED DESCRIPTION:
This study is divided into two parts. Part A is a multicenter, randomized, double-blind, placebo controlled phase Ill clinical trial, designed to evaluate the efficacy and safety of ZM-H1505R in combination with NAs versus NAs monotherapy with HBV DNA ≥ 50 IU/mL and are HBeAg positive who have received NAs monotherapy for at least 12months.Part B is an open-label extension and follow-up period designed to evaluate the long-term safety and efficacy of ZM-H1505R in combination with NAs.

- Part A (Double-Blind Treatment Period): Eligible subjects will be randomized in a 1:1 ratio into 2 groups. Group A:ZM-H1505R 100mg +NAs Group B:ZM-H1505R placebo +NAs Two randomization stratification factors were set: NAs type of ETV, TDF,TAF, or TMF (no less than 15% of ETV, TDF, and TAF); HBV DNA <2000 IU/mL and HBV DNA >2000 IU/mL . All subjects completed a 48-week efficacy and safety evaluation followed by an interim analysis, the results of which were used to submit an NDA application.

- Part B (Open-Label Extension Period): At the end of the 48-week randomized double-blind treatment period, all eligible subjects will transfer to the open-label extension period and were treated with ZM-H1505R 100 mg +NAs while the study drug was evaluated for efficacy and safety until the end of the 144 weeks.

- Follow-up Period: At the end of the 144-week open-label extension period, all subjects will continue to take NAs, as a monotherapy for a 4-week follow-up period for observation of efficacy and safety of after discontinuation of study drug in ZM-H1505R .

ELIGIBILITY:
Inclusion Criteria:

* 1.Able to understand and sign the written informed consent form;
* 2.Adult males and females aged 18-65 years(inclusive) at screening;
* 3.Have been used NAs monotherapy with ETV(0.5 mg or 1.0mg, QD),TDF (300 mg, QD),TAF (25 mg, QD),or TMF (25 mg, OD)for at least 12 months at the time of enrollment; Have been on stable and continuous use of one of these medications for at least 6months, and do not plan to switch to any other NAs class of medications after entering this clinical trial;
* 4.Evidence of prior HBV infection (e.g., HBsAg and/or HBV DNA positive), or HBsAg positive at screening;
* 5.HBV DNA ≥50 IU/mL as measured by a local healthcare facility within 30 days prior to screening and HBV DNA ≥50 IU/mL as confirmed by central laboratory testing at the time of screening;
* 6.HBeAg positivity confirmed by central laboratory testing at screening;
* 7.Women of childbearing potential or males with female partners of childbearing potential must agree to voluntarily use the contraceptive methods specified in the protocol from screening to 28 days after the last dose of the study.

Exclusion Criteria:

* 1.Progressive fibrosis or cirrhosis detected at screening, or progressive fibrosis or cirrhosis defined as follows: Metavir ≥ 3 or Ishak fibrosis score ≥ 4 by liver biopsy within 1 year prior to screening; or in the absence of an appropriate liver biopsy, liver stiffness test (FibroScan) ≥ 9 kPa within 3 months prior to screening, or liver stiffness test (FibroTouch) ≥ 9.6 kPa(FibroScan preferred) ;
* 2.History of hepatocellular carcinoma (HCC); or serum alpha-fetoprotein (AFP) ≥ 50 ng/mL at screening, or imaging examination such as abdominal ultrasound, CT (computed tomography) or MRI (magnetic resonance imaging) suggesting possible HCC;
* 3.Subjects meeting any of the following clinical laboratory parameters at screening:

  1. Hemoglobin < 110 g/L (for males) or < 100 g/L (for females);
  2. Platelet count < 90 × 109/L;
  3. Neutrophil count < 1.5 × 109/L;
  4. Alanine aminotransferase (ALT) or Aspartate aminotransferase(AST)> 3 × upper limit of normal (×ULN);
  5. International normalized ratio (INR) of prothrombin time > 1.3;
  6. Albumin < 35 g/L;
  7. Total bilirubin > 2 × ULN, and direct bilirubin > 1.5 × ULN;
  8. Estimated glomerular filtration rate < 60 mL/min/1.73 m2(calculated using the CKD-MDRD formula).
* 4.Abnormal result of electrocardiogram (ECG) at screening and inappropriate for the study participation judged by the investigator; or QTcF (QT corrected using the Fridericia formula): > 450 ms for males, > 470 ms for females at screening;
* 5.Co-infection with human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV) or hepatitis E virus (HEV); Note: Subjects with positive HCV antibody (Ab) but negative HCV RNA and subjects with positive HEV immunoglobulin M (IgM) but negative HEV RNA will NOT be excluded.
* 6.Other malignancy unless the subject's malignancy has been cured by surgical resection (e.g., basal cell skin cancer); Note: Subjects who are suspected of having malignancy must be excluded regardless of evidence of local recurrence or metastasis.
* 7.History of chronic liver disease with a non-HBV etiology, such as alcoholic liver disease, autoimmune liver disease, hereditary liver disease, non-alcoholic fatty liver disease, except for simple fatty liver disease;
* 8.Other concurrent severe systemic diseases or clinical manifestations, for which the investigator considers not suitable to participate in this study;
* 9.Use of any investigational product or drug not approved by regulatory authorities within 3 months prior to screening;
* 10.History of persistent alcohol consumption (alcohol consumption exceeding 40 g ethanol for males or 20g ethanol for females per day on average) within 6 months prior to screening;
* 11.History of drug dependence or drug abuse;
* 12.Pregnant or breastfeeding women;
* 13.Known hypersensitivity to the active ingredient or formulation excipients of the investigational drug;
* 14.Inappropriate for the study participation for any reason not otherwise listed as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieves complete virologic response (CVR) at week 48 of treatment. | 48 week
  To evaluate the efficacy of ZM-H1505R in combination with NAs versus NAs monotherapy in adult CHB subjects who have received NAs monotherapy for at least 12 months. (CVR is defined as HBV DNA ≤ 10 IU/mL)

SECONDARY OUTCOMES:
Safety of ZM-H1505R in combination with NAs versus NAs monotherapy in adult CHB subjects who have received NAs monotherapy for at least 12 months. | From baseline to the end of follow-up period(Part A and Part B), assessed up to 148 weeks.
  Safety during the 48-week double-blind treatment period, the open-label extension period, and the follow-up period.
Percentage of subjects who achieve CVR at each scheduled visit other than week 48 visit | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
  CVR is defined as HBV DNA ≤ 10 IU/mL).
Time to achieve CVR in each group | Part A(double-blind treatment period):from baseline to week 48
  CVR is defined as HBV DNA ≤ 10 IU/mL
Percentage of subjects with quantitative HBV DNA ≤ 20 IU/mL | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
Changes from baseline in quantitative HBV RNA | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
Percentage of subjects who achieve LLOQ of quantitative HBV RNA | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
Changes from baseline in quantitative serum HBsAg | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
Changes from baseline in HBeAg at each scheduled visit | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
Changes from baseline in quantitative serum HBcrAg at each scheduled visit; | Part A(double-blind treatment period):from baseline to week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.
Changes from baseline in liver stiffness test (FibroScan/FibroTouch) | Part A(double-blind treatment period):at week24 and week 48; Part B (open-label extension period and follow-up period):from week 48 to week 148.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No